CLINICAL TRIAL: NCT06945172
Title: Comparison of Prostate Cancer-related Quality of Life in Sexually Active Men With Favourable Intermediate-risk Localised Prostate Cancer Treated With Total Prostatectomy or Focal HIFU
Acronym: QUALIFY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-A02716-41; 2024-A02716-41 (Other: ANSM)
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total prostatectomy (Active Comparator): Patient will undergo total prostatectomy as a treatment for their cancer
  Interventions: Procedure: Total prostatectomy
- Focal HIFU (Experimental): Patient will undergo focal HIFU as a treatment for their cancer
  Interventions: Procedure: Focal HIFU

INTERVENTIONS:
Procedure: Total prostatectomy — Total prostatectomy is a surgical procedure performed to treat prostate cancer.
  Arms: Total prostatectomy
Procedure: Focal HIFU — Focal HIFU treatment is an innovative technique that consists of destroying prostate tumour cells using high-intensity ultrasound focused exclusively on the affected area of the gland.
  Arms: Focal HIFU

SUMMARY:
The goal of this trial is to assess the impact of focal HIFU therapy on quality of life in patients with favourable intermediate-risk localised prostate cancer. The main question it aims to answer is:

What is the prostate cancer-related quality of life in patients with favourable intermediate-risk localised cancer treated by total prostatectomy or focal HIFU ?

Researchers will compare patients with favourable intermediate-risk localised cancer treated by total prostatectomy to patients with favourable intermediate-risk localised cancer treated by focal HIFU to see their quality of life.

Participants will answer EPIC-CP questionnaire 6 months, 12 months and 24 months after treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient, male, aged between ≥ 40 and ≤ 75 years
* Patient with a life expectancy > 10 years at the time of inclusion.
* Patient with a therapeutic strategy (prostatectomy or focal HIFU) defined during a PCR.
* Patient with a diagnosis of localised prostate cancer at favourable intermediate risk
* Patient able to tolerate general anaesthesia or type IV sedation
* Patient with normal urinary continence status
* Patient with satisfactory erectile function allowing penetration:
* Patient with targeted biopsies and systematic biopsies
* Patient affiliated to or benefiting from a social security scheme
* French-speaking patients who do not object to the use of their data.

Exclusion Criteria:

* Patients with a contraindication to MRI
* Stage T3a or b on MRI
* Patient on long-term anticoagulants and unable to stop them.
* Patient already included in another study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study deals with prostate cancer so that only men are eligible to participate
Enrollment: 102 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in relation to prostate cancer | Month 6, month 12 and month 24
  Quality of life in relation to prostate cancer will be assessed by the total score (ranging from 0 to 60) of the EPIC-CP (Expanded Prostate Cancer Index Composite for Clinical Practice) questionnaire. Higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique La Croix du Sud, Quint-Fonsegrives, France